CLINICAL TRIAL: NCT03396614
Title: Detection of (Sub)Clinical Toxicity in Irradiated vs. Non-irradiated Surgically Treated Esophageal Cancer Patients: a Pilot Study (CROSS SECT)
Acronym: CROSS SECT
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2017-06/ METc 2017/335
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Thoracic Tumor
MeSH Terms: conditions — Thoracic Neoplasms | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EEG, ECG, CT, MRI
  Interventions: Diagnostic Test: CTTC scan, cardiac MRI, ECG, 6 minute walking test, echocardiogram

INTERVENTIONS:
Diagnostic Test: CTTC scan, cardiac MRI, ECG, 6 minute walking test, echocardiogram — CTTC scan, cardiac MRI, ECG, 6 minute walking test, echocardiogram

SUMMARY:
Rationale: Radiation-induced cardiac and pulmonary toxicity after treatment for intra-thoracic tumors is a clinically relevant problem, which may jeopardize the benefit of (neo-adjuvant) (chemo) radiotherapy. Although cure rates are rising since the introduction of neo-adjuvant chemoradiation (neo-CRT) as current standard treatment for esophageal cancer (EC), recent studies showed that there is a substantial risk of non-cancer treatment-related death in these patients. Furthermore, this risk is underestimated as the cause of death of many patients remains unknown, since the distinction between tumor related and non-cancer related death can be difficult.

Cardiac and pulmonary toxicity and its interaction as seen in pre-clinical studies might explain for these unknown deaths as suggested in several clinical studies. Clinical imaging studies performed shortly after treatment showed changes in different cardiac function parameters, all related to radiation dose parameters. Systematic imaging studies analysing subclinical toxicities at longer follow up have never been performed, most probably because of poor survival rates. However, identification of the magnitude of (subclinical) cardiopulmonary toxicity, by performing several cardiopulmonary function tests, is essential in this patient group as this toxicity is most likely the cause of the increased mortality after thoracic radiotherapy. For future perspectives, these results can be used to select the best diagnostic methods for a prospective cohort study to develop prediction tools for cardiopulmonary toxicity..

Objective: The main objective of this study is to determine the most suitable diagnostic test to identify cardiopulmonary (dys)function in EC survivors treated with neo-CRT followed by surgical resection. Furthermore, we want to estimate the difference in cardiopulmonary (dys)function in EC survivors treated with neo-CRT followed by surgical resection compared to EC survivors who were treated with surgical resection alone.

Study design: Cross-sectional pilot study

Study population: 40 EC patients who were treated with curative intent by esophageal resection with or without neo-CRT

Intervention (if applicable): Not applicable.

Main study parameters/endpoints: As this is an exploratory pilot study to determine the most suitable diagnostic tests for future studies, there will be several endpoints related to (sub)clinical cardiopulmonary dysfunction.

Signs of myocardial ischemia, systolic or diastolic dysfunction, rhythm and valve disorders, pericardial effusion and fibrosis, myocardial fibrosis, focal wall motion disorders and coronary calcifications will be analyzed. The cardiopulmonary (dys)function in EC survivors treated with neo-CRT followed by surgical resection will be compared to cardiopulmonary (dys)function in EC survivors treated with surgical resection alone.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Several tests will be performed at one time point, 5-10 years after given treatment. If the findings of the test indicate cardiovascular complications, the patient will be referred to the cardiologist for further analysis and/or preventive measures. As one of the tests, cardiac MRI, including gadolinium (Dotarem 0.2 mmol/kg) enhancement will be performed. Potential side effects of gadolinium include brief headache, nausea (feeling sick) and dizziness for a brief time following the injection. Allergic reactions are rare. Furthermore, a cardiac CT scan will be performed with a total radiation exposure of 0.6 mSv (less than a third of the annual background radiation dose), the risks will be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Treated for EC with a curative resection between 2000 and 2012
* Age >= 18 years
* Written informed consent
* No signs of tumor recurrence or new other malignancies.

Exclusion Criteria:

* Thoracic radiotherapy for indications other than EC.
* Contra indication for cardiac MRI, pacemaker, cochlear implants, metal not compliable with MRI.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EC treated with or without neo-CRT, alive without evidence of disease, treated between 2000 and 2012 at the University Medical Centre Groningen will be eligible. Twenty patients will be included in both treatment groups. Length of follow up after treatment does not seem to be an important confounding factor as surgery is not considered to be an important risk factor for late toxicity.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The cardiopulmonary (dys)function in EC survivors treated with neo-CRT followed by surgical resection will be compared to cardiopulmonary (dys)function in EC survivors treated with surgical resection alone. | cross sectional 5-10 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Beukema, Dr., Principal Investigator — Radiation oncologist
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03396614/Prot_000.pdf